CLINICAL TRIAL: NCT05356884
Title: An Adolescent-mediated Intervention to Improve Diabetes Prevention and Management in Pacific Islander Families
Brief Title: Adolescent-mediated Family Diabetes Intervention: American Samoa
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000031325; 1R01DK128277-01A1 (NIH)
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus; American Samoa; Adolescent; Pacific Islander
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Leadership

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes Intervention (Experimental): 12-session behavioral intervention covering diabetes pathology, self-monitoring, medication adherence, identifying and responding to emergency situations, diet, physical activity, health care utilization and maintaining healthy habits.
  Interventions: Behavioral: Diabetes Intervention
- Leadership & Life Skills (Active Comparator): 12-session leadership and life skills intervention focusing on adolescent self-esteem, self-efficacy, communication skills, mindfulnesss, healthy habits.
  Interventions: Behavioral: Leadership & Life Skills

INTERVENTIONS:
Behavioral: Diabetes Intervention — A 12-session group-based intervention that will target diabetes knowledge and leadership and communication skills through facilitated discussion and experiential learning.
  Arms: Diabetes Intervention
Behavioral: Leadership & Life Skills — A 12-session group based intervention that will teach leadership and life skills (planning strategies, leadership values, emotional awareness, effective reasoning skills)
  Arms: Leadership & Life Skills

SUMMARY:
The goal of this project is to test the feasibility, acceptability, and preliminary efficacy of an adolescent-mediated intervention designed to improve the glycemic control and self-care practices of a parent/grandparent. The preliminary impact of the intervention on adult glycemic control (HbA1c) and self-care behaviors, as well as adolescent risk factors, will be explored with the goal of informing future programs that can be scaled to reduce diabetes burden and eliminate health disparities among at risk, ethnic minority groups.

DETAILED DESCRIPTION:
The number of individuals diagnosed with Type 2 Diabetes in the United States (US) has more than doubled since 2000 to over 30 million, with an additional 84.1 million living with prediabetes. One minority group at particular risk is Pacific Islanders (PIs), who are at disproportionate risk and face many barriers (structural and cultural) to engaging in prevention or self-care. To address the critical need for diabetes prevention and treatment programs that target PIs, and building on the family-centered culture, the objective of this project is to pilot test and evaluate a randomized controlled trial of an adolescent-mediated intervention designed to improve the glycemic control and self-care practices of a paired, adult family member with diagnosed diabetes. Dyads (n=160 dyads; an adolescent without diabetes and a parent/grandparent diagnosed with diabetes who share a household) will be randomized. Adolescents will receive either a six-month diabetes intervention or a leadership and life skills-focused control curriculum in groups (n=10 participants in each group). Aside from planned research assessments there will be no contact with the adults in the dyad, who will proceed with their usual diabetes care. To test the hypothesis that adolescents receiving the intervention will be effective conduits of diabetes knowledge and will support their paired adult in the adoption of self-care strategies, the primary efficacy outcomes will be adult glycemic control and cardiovascular risk factors (BMI, blood pressure, waist circumference). Secondarily, since exposure to the intervention may encourage positive behavior change in the adolescent themselves similar outcomes will be measured in the adolescents. Outcomes will be measured at baseline, at the end of the active intervention phase (six months post-randomization) and at 12-months post-randomization, to examine maintenance of intervention effects in the absence of contact. To determine potential for long-term sustainability and scale up, program acceptability, feasibility, fidelity, reach, and cost will be examined. Successful completion of the study aims and proof of efficacy would produce an innovative, scalable program with high potential for replication in other similar, low-resource, family-centered, ethnic minority groups across the US who are the ideal beneficiaries of innovations to reduce chronic disease risk and eliminate health disparities.

ELIGIBILITY:
Inclusion Criteria:

Adolescent

* 14-17 years of age
* Samoan ethnicity
* Shares a household with a parent, legal guardian, or grandparent with type II diabetes
* Willing and able to consent to participation
* Able to participate in group sessions after school or on Saturday mornings

Adult

* Samoan ethnicity
* Diagnosed with type II diabetes at least 12 months prior to study enrollment
* HbA1c >= 6.5%
* Prescribed medication (tablets or insulin) to control their diabetes
* Willing and able to consent to participation
* Willing and able to consent to adolescent's participation

Exclusion Criteria:

Adolescent

* Planning to become pregnant during the study period (any adolescent who becomes pregnant will be excluded from analysis)
* Planning to leave American Samoa in the next 18 months
* Participants will be excluded if they report any of the following:

  * Uncontrolled hypertension (systolic >180 mmHg or diastolic >105 mmHg)
  * Heart attack, stroke, or transient ischemic attack in the past year
  * Treatment for cancer
  * Chest pain or shortness of breath with minimal activity
  * Chronic lung disease, or asthma requiring home oxygen therapy
  * Contraindications to moderate physical activity
  * Inability to read/speak Samoan and/or English.
* Overt diabetes (HbA1c ≥6.5%) based on point-of-care testing during the screening process

Adult

* Planning to become pregnant during the study period (any adult who becomes pregnant will be excluded from analysis)
* Planning to leave American Samoa in the next 18 months
* Participants will be excluded if they report any of the following:

  * Uncontrolled hypertension (systolic >180 mmHg or diastolic >105 mmHg)
  * Heart attack, stroke, or transient ischemic attack in the past year
  * Treatment for cancer
  * Chest pain or shortness of breath with minimal activity
  * Chronic lung disease, or asthma requiring home oxygen therapy
  * Contraindications to moderate physical activity
  * Inability to read/speak Samoan and/or English.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Adult Glycemic Control (HbA1c) 0-6 months | 0 - 6 months
  Glycated hemoglobin (marker of long term glycemic control)
Change in Adult Glycemic Control (HbA1c) 0-12 months | 0 - 12 months
  Glycated hemoglobin (marker of long term glycemic control)
Change in Adult Glycemic Control (HbA1c) 6-12 months | 6 - 12 months
  Glycated hemoglobin (marker of long term glycemic control)
Change in Adult Body Mass Index (BMI) 0-6 months | 0 - 6 months
  Body mass index (measure of weight control)
Change in Adult Body Mass Index (BMI) 0-12 months | 0 - 12 months
  Body mass index (measure of weight control)
Change in Adult Body Mass Index (BMI) 6-12 months | 6 - 12 months
  Body mass index (measure of weight control)
Change in Adult Blood Pressure (BP) 0 - 6 months | 0 - 6 months
  Blood Pressure (marker of hypertension risk)
Change in Adult Blood Pressure (BP) 0 - 12 months | 0 - 12 months
  Blood Pressure (marker of hypertension risk)
Change in Adult Blood Pressure (BP) 6 - 12 months | 6 - 12 months
  Blood Pressure (marker of hypertension risk)
Change in Adult Waist Circumference (WC) 0 - 6 months | 0 - 6 months
  Waist circumference (measure of weight control)
Change in Adult Waist Circumference (WC) 0 - 12 months | 0 - 12 months
  Waist circumference (measure of weight control)
Change in Adult Waist Circumference (WC) 6 - 12 months | 6 - 12 months
  Waist circumference (measure of weight control)

SECONDARY OUTCOMES:
Change in Adolescent Glycemic Control (HbA1c) 0 - 6 months | 0 - 6 months
  Glycated hemoglobin (marker of long term glycemic control)
Change in Adolescent Glycemic Control (HbA1c) 0 - 12 months | 0 - 12 months
  Glycated hemoglobin (marker of long term glycemic control)
Change in Adolescent Glycemic Control (HbA1c) 6 - 12 months | 6 - 12 months
  Glycated hemoglobin (marker of long term glycemic control)
Change in Adolescent Body Mass Index (BMI) 0 - 6 months | 0 - 6 months
  Body mass index (measure of weight control)
Change in Adolescent Body Mass Index (BMI) 0 - 12 months | 0 - 12 months
  Body mass index (measure of weight control)
Change in Adolescent Body Mass Index (BMI) 6 - 12 months | 6 - 12 months
  Body mass index (measure of weight control)
Change in Adolescent Blood Pressure (BP) 0 - 6 months | 0 - 6 months
  Blood Pressure (marker of hypertension risk)
Change in Adolescent Blood Pressure (BP) 0 - 12 months | 0 - 12 months
  Blood Pressure (marker of hypertension risk)
Change in Adolescent Blood Pressure (BP) 6 - 12 months | 6 - 12 months
  Blood Pressure (marker of hypertension risk)
Change in Adolescent Waist Circumference (WC) 0 - 6 months | 0 - 6 months
  Waist circumference (measure of weight control)
Change in Adolescent Waist Circumference (WC) 0 - 12 months | 0 - 12 months
  Waist circumference (measure of weight control)
Change in Adolescent Waist Circumference (WC) 6 - 12 months | 6 - 12 months
  Waist circumference (measure of weight control)

CONTACTS AND LOCATIONS:
Overall Officials: Nicola L Hawley, PhD, Principal Investigator — Yale University School of Public Health
Locations (1):
- OLaGA Research Center, Pago Pago, American Samoa

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with other researchers for the purpose of analyses agreed upon with the Principal Investigator
Supporting Information: Study Protocol, SAP
Time Frame: Study protocol has been published and is available at: https://journals.plos.org/plosone/article?id=10.1371/journal.pone.0279084
  Detailed intervention and control curricula will be available in August 2024 upon completion of data collection.
Access Criteria: All materials will be made publicly available.
URL: https://journals.plos.org/plosone/article?id=10.1371/journal.pone.0279084

REFERENCES:
- [Derived] Hawley NL, Rivara AC, Naseri J, Faumuina K, Potoa'e-Solaita N, Iopu F, Faiai M, Naveno E, Tasele S, Lefale T, Lantini R, Carlson JC, Rabin TL, Semaia P, Mugadza P, Rosen RK. Protocol: Implementation and evaluation of an adolescent-mediated intervention to improve glycemic control and diabetes self-management among Samoan adults. PLoS One. 2023 Feb 16;18(2):e0279084. doi: 10.1371/journal.pone.0279084. eCollection 2023. PMID 36795707

DOCUMENTS (1):
  • Informed Consent Form (2022-02-25): https://cdn.clinicaltrials.gov/large-docs/84/NCT05356884/ICF_000.pdf